CLINICAL TRIAL: NCT06800261
Title: A Randomized, Double-blind, Positive Controlled Phase Ib Clinical Trial to Evaluate the Safety and Immunogenicity of 24-valent Pneumococcal Conjugate Vaccine in Children Aged 2 (Minimum 42 Days)-23 Months
Brief Title: Clinical Trial of PCV24 in Infants Aged 2-23 Months
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-PCV24-1003
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Sinovac PCV24 (Experimental): Participants aged 2 months (minimum 42 days)-23 months will receive Sinovac PCV24 according to different immunization schedules. Route of administration is intramuscular injection at anterolateral thigh for infants aged younger than 12 months, and at deltoid muscle of upper arm for children aged older than 12 months.
  Interventions: Biological: Sinovac PCV24
- Active Comparator: Prevnar® (Active Comparator): Participants aged 2 months (minimum 42 days)-23 months will receive Prevnar 13® according to different immunization schedules. Route of administration is intramuscular injection at anterolateral thigh for infants aged younger than 12 months, and at deltoid muscle of upper arm for children aged older than 12 months.
  Interventions: Biological: Prevnar®

INTERVENTIONS:
Biological: Sinovac PCV24 — Sinovac PCV24 (0.5 mL) is administered intramuscularly according to different immunization schedules.
  Arms: Experimental: Sinovac PCV24
Biological: Prevnar® — Prevnar® (0.5 mL) is administered intramuscularly according to different immunization schedules.
  Arms: Active Comparator: Prevnar®

SUMMARY:
A Phase 1b clinical trial of 24-valent pneumococcal conjugate vaccine (PCV24) developed by Sinovac Life Science Co., Ltd will be conducted in pediatric population aged 2 months (minimum 42 days)-23 months.

The objective of the study is to evaluate the safety and immunogenicity of Sinovac PCV24. The trial is a randomized, double-blind, positive controlled phase Ib clinical trial.

DETAILED DESCRIPTION:
A phase 1b clinical trial of the study of 24-valent Pneumococcal Polysaccharide Conjugate Vaccine (PCV24) developed by Sinovac Life Science Co., Ltd (Sinovac) will be conducted in Chinese pediatric population aged 2 months (minimum 42 days)-23 months. The trial is a randomized, double-blind, positive controlled study. The objective of this study is to evaluate the safety and immunogenicity of PCV24 manufactured by Sinovac Life Science Co., Ltd. The active control vaccine is Prevenar13® manufactured by Pfizer.

A total of at least 180 participants aged 2 months (minimum 42 days)-23 months will be enrolled. Participants will be randomized in 1:1 ratio to the test group and control group.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants who are aged 2 months (42-89 days), 7-11 months, 12-23 months;
2. Participants' guardian provides legal identity document and participants' vaccination record;
3. Participants' guardian understands and voluntarily signs the informed consent form;
4. Follow all study procedures and stay in contact during the study.

Exclusion Criteria:

1. Received any pneumococcal vaccine prior to enrollment;
2. History of invasive pneumococcal diseases or other pneumococcal diseases caused by Streptococcus pneumoniae, as confirmed by laboratory tests;
3. History of severe adverse reactions to the vaccine or vaccine components, or history of allergy, such as urticaria, dyspnea, angioneurotic edema, anaphylactic shock;
4. Low birth weight (<2.5kg), or premature infant (gestation weeks < 37 weeks) (applies to infants younger than 12 months);
5. History of abnormal labor during delivery (planned cesarean section is excluded), history of asphyxia rescue and nervous system damage (applies to infants younger than 12 months);
6. Congenital malformations or developmental disorders, genetic defects, severe malnutrition;
7. Have uncontrolled chronic diseases or history of severe diseases, including but not limited to cardiovascular diseases (e.g. congenital heart disease), hematological diseases (e.g. severe anemia), liver and kidney diseases, digestive diseases, respiratory diseases (such as active tuberculosis), malignant tumors and major functional organ transplantation history;
8. Autoimmune diseases, immunodeficiency diseases (including but not limited to systemic lupus erythematosus, rheumatoid arthritis, autoimmune thyroid disease, asplenia, functional asplenia, HIV infection);
9. Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets level), potential bleeding (history of obvious bleeding, hematoma or bruising after intramuscular injection or venipuncture).
10. Have/have suffered from a serious neurological disorder (epilepsy or convulsions, but febrile convulsion is not an exclusion criteria ) or mental illness or have a family history of such diseases.
11. Consecutively received immunosuppressive therapy (excluding corticosteroid spray therapy for allergic rhinitis and surface corticosteroid therapy for acute non-concurrent dermatitis), or other immunoregulatory therapies, or cytotoxic therapy over 14 days within 6 months before vaccination, or plans to receive such therapies during the study.
12. Received blood products prior to enrollment within 3 months prior to enrollment, or plans to receive such therapies during the study. Receipt of Hepatitis B immunoglobulin one month prior to enrollment is an exception.
13. Received other investigational drugs or vaccines within 30 days prior to enrollment, or plan to receive such drugs or vaccines during the study;
14. Received live attenuated vaccine within 14 days prior to enrollment;
15. Received subunit or inactivated vaccine within 7 days prior to enrollment;
16. Acute diseases or acute onset of chronic diseases within 7 days prior to enrollment, known or potentially active infection;
17. Axillary temperature≥ 37.3 Degree Celsius before vaccination;
18. In the investigator's judgment, the participant has any other factors that make him or her unfit to participate in the clinical trial.

Ages: 42 Days to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions | 0-30 days after vaccination
  Incidence of adverse reactions within 30 days after vaccination

SECONDARY OUTCOMES:
Incidence of adverse reactions | 0-7 days after vaccination
  Incidence of adverse reactions within 7 days after vaccination
Incidence of serious adverse events (SAE) | from vaccination to 6 months after final dose
  Incidence of SAE during the period of safety monitoring
Pneumococcal serotype-specific IgG antibody geometric mean concentration (GMC) | 30 days after primary vaccination
  IgG GMC 30 days after primary vaccination
Pneumococcal serotype-specific IgG antibody geometric mean increase (GMI) | 30 days after primary vaccination
  IgG GMI 30 days after primary vaccination
Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 1.0 μg/mL | 30 days after primary vaccination
  Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 1.0 μg/mL
Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 0.35 μg/mL (seropositive rate) | 30 days after primary vaccination
  Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 0.35 μg/mL (seropositive rate)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Xu, Principal Investigator — Shandong Provincial Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Shandong Provincial Center for Disease Control and Prevention, Jinan, Shandong
  - Shanxian Center for Disease Control and Prevention, Shancheng, Shandong